CLINICAL TRIAL: NCT00240526
Title: Comparative Study of the Immunogenicity and Protective Efficacy of GlaxoSmithKline Biologicals' Rec-DNA Hepatitis B Vaccine With or Without Hepatitis B Immunoglobulins (HBIg) in Newborns of HBeAg+ Mothers.
Brief Title: LT F-up Study 16-20 Yrs After Vaccine Dose of Hepatitis B With/Without HBIg in Newborns to HBeAg+ Mothers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100450
Record Dates: First submitted 2005-10-13; First posted 2005-10-18 (Estimated); Results first posted 2010-07-15 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis B immunoglobulin; Hepatitis B antibody persistence
MeSH Terms: conditions — Hepatitis B | interventions — hepatitis B hyperimmune globulin

ARMS (4):
- Engerix 4D + HBIg Group (Experimental): Subjects received Engerix™ (hepatitis B vaccine [HBV]) at Month 0, 1, 6 and 60 with hepatitis B immunoglobulins (HBIg) administered concomitantly at birth in the opposite arm.
  Interventions: Biological: Engerix™ -B; Biological: Hepatitis B immunoglobulin (HBIg)
- Engerix 3D + HBIg Group (Experimental): Subjects received Engerix™ (hepatitis B vaccine [HBV]) at Month 0, 1, and 6 with hepatitis B immunoglobulins (HBIg) administered concomitantly at birth in the opposite arm.
  Interventions: Biological: Engerix™ -B; Biological: Hepatitis B immunoglobulin (HBIg)
- Engerix 4D (Experimental): Subjects received Engerix™ (hepatitis B vaccine [HBV]) at Month 0, 1, 6 and 60.
  Interventions: Biological: Engerix™ -B
- Engerix 3D Group (Experimental): Subjects received Engerix™ (hepatitis B vaccine [HBV]) at Month 0, 1, and 6.
  Interventions: Biological: Engerix™ -B

INTERVENTIONS:
Biological: Engerix™ -B — 3 (Groups A and C) or 4 (Groups B and D) intramuscular injections during the primary study
Biological: Hepatitis B immunoglobulin (HBIg) — 1 intramuscular injections at birth (primary study)
  Arms: Engerix 3D + HBIg Group; Engerix 4D + HBIg Group

SUMMARY:
To evaluate the persistence of anti-HBs antibodies up to 16, 17, 18, 19 and 20 years after administration of the first dose of the study vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

No additional subjects will be recruited during this long-term follow-up study and no vaccine will be administered.

DETAILED DESCRIPTION:
The primary study was to evaluate the reactogenicity, immunogenicity and protective efficacy of a hepatitis B vaccine in healthy neonates of HBeAg positive mothers if administered with or without a dose of HBIg at birth. The current study describes the long term follow up of these subjects between Y16 and 20 after primary vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had received at least one dose of the study vaccine in the primary study
* Written informed consent obtained from each subject before each blood sampling visit

Exclusion Criteria:

* None

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2003-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Leroux-Roels G, Crasta PD, Hardt K. Persistence and immune memory to hepatitis B vaccine 20 years after primary vaccination of Thai infants, born to HBsAg and HBeAg positive mothers. Hum Vaccin Immunother. 2012 Jul;8(7):896-904. doi: 10.4161/hv.19989. Epub 2012 Jul 1. PMID 22777097
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The baseline characteristics are given for the Year 15 time point. Therefore the number of participants in the Engerix-3D Group is 21, as in the Year 15 participant flow data.
Period: Year 15
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 19 (Number of subjects who come back at Year 15 (Month 180) time-point) | 19 (Number of subjects who come back at Year 15 (Month 180) time-point) | 14 (Number of subjects who come back at Year 15 (Month 180) time-point) | 21 (Number of subjects who come back at Year 15 (Month 180) time-point)
Completed | 19 | 19 | 14 | 21
Not Completed | 0 | 0 | 0 | 0
Period: Year 16
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 17 (Number of subjects who come back at Year 16 (Month 192) time-point) | 19 (Number of subjects who come back at Year 16 (Month 192) time-point) | 16 (Number of subjects who come back at Year 16 (Month 192) time-point) | 22 (Number of subjects who come back at Year 16 (Month 192) time-point)
Completed | 17 | 19 | 16 | 22
Not Completed | 0 | 0 | 0 | 0
Period: Year 17
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 19 (Number of subjects who come back at Year 17 (Month 204) time-point) | 17 (Number of subjects who come back at Year 17 (Month 204) time-point) | 13 (Number of subjects who come back at Year 17 (Month 204) time-point) | 20 (Number of subjects who come back at Year 17 (Month 204) time-point)
Completed | 19 | 17 | 13 | 20
Not Completed | 0 | 0 | 0 | 0
Period: Year 18
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 16 (Number of subjects who come back at Year 18 (Month 216) time-point) | 17 (Number of subjects who come back at Year 18 (Month 216) time-point) | 14 (Number of subjects who come back at Year 18 (Month 216) time-point) | 20 (Number of subjects who come back at Year 18 (Month 216) time-point)
Completed | 16 | 17 | 14 | 20
Not Completed | 0 | 0 | 0 | 0
Period: Year 19
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 17 (Number of subjects who come back at Year 19 (Month 228) time-point) | 16 (Number of subjects who come back at Year 19 (Month 228) time-point) | 12 (Number of subjects who come back at Year 19 (Month 228) time-point) | 18 (Number of subjects who come back at Year 19 (Month 228) time-point)
Completed | 17 | 16 | 12 | 18
Not Completed | 0 | 0 | 0 | 0
Period: Year 20
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Started | 19 (Number of subjects who come back at Year 20 (Month 240) time-point) | 17 (Number of subjects who come back at Year 20 (Month 240) time-point) | 13 (Number of subjects who come back at Year 20 (Month 240) time-point) | 20 (Number of subjects who come back at Year 20 (Month 240) time-point)
Completed | 19 | 17 | 13 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group | Total
Number analyzed (Participants) | 19 | 19 | 14 | 21 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] — Data are given for the Year 15 time point.
  years | 14.5 (0.51) | 14.7 (0.45) | 14.6 (0.50) | 14.5 (0.51) | 14.6 (0.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 6 | 10 | 35
  Male | 7 | 12 | 8 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration as Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Description: Concentrations given as GMC expressed as milli-international unit per millilitre (mIU/mL).
  Note: At Year 15 and 16, a commercial ELISA was used. From Year 17 to Year 20, anti-HBs antibody concentrations were tested with a validated in-house assay with cut-off 3.3mIU/mL.
Time Frame: At Years 15, 16, 17, 18, 19 and 20
Population: Analysis was performed on subjects from the Long Term According-to-Protocol (LT ATP) cohort for immunogenicity on subjects with available data at the specified time-points
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Number analyzed (Participants) | 17 | 15 | 12 | 17
mIU/mL
  Year 15 (N=17;15;12;17) | 118.6 [53.4 to 263.1] | 14.8 [6.8 to 32.0] | 142.8 [30.4 to 669.4] | 24.2 [10.0 to 58.7]
  Year 16 (N=15;13;12;16) | 119.3 [50.0 to 284.7] | 14.1 [6.8 to 29.4] | 134.3 [30.1 to 599.8] | 22.9 [9.7 to 54.1]
  Year 17 (N=17;13;11;13) | 140.0 [67.2 to 291.9] | 8.2 [3.9 to 17.1] | 70.2 [14.3 to 344.1] | 17.0 [6.7 to 43.3]
  Year 18 (N=14;14;10;13) | 82.3 [32.1 to 211.3] | 10.8 [6.5 to 17.9] | 56.5 [11.7 to 271.8] | 26.1 [10.7 to 63.3]
  Year 19 (N=13;12;8;11) | 103.3 [38.9 to 274.7] | 9.5 [4.0 to 22.8] | 84.9 [12.0 to 600.2] | 19.9 [7.4 to 53.7]
  Year 20 (N=13;13;6;12) | 73.9 [26.6 to 205.4] | 14.3 [6.7 to 30.6] | 297.1 [46.0 to 1919.5] | 16.3 [7.2 to 36.9]

2. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration as Measured by ChemiLuminescence ImmunoAssay (CLIA).
Description: Concentrations given as GMC expressed as milli-international unit per millilitre (mIU/mL).
  Note: There was a change of assay kit at Year 19 time-point, thus for the sake of bridging, blood samples corresponding to Year 19 were re-tested with new CLIA. At Year 19 and 20, anti-HBs antibody concentrations tested with the CLIA with cut-off 6.2 mIU/mL.
Time Frame: At Years 19 and 20
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | ENGERIX 4D + HBIG GROUP | ENGERIX 3D + HBIG GROUP | ENGERIX 4D | ENGERIX 3D GROUP
Number analyzed (Participants) | 16 | 13 | 7 | 13
mIU/mL
  YEAR 19 (N=14;12;6;11) | 60.1 [26.7 to 135.5] | 5.8 [3.3 to 10.0] | 159.0 [32.6 to 776.5] | 11.7 [5.0 to 27.4]
  YEAR 20 (N=16;13;7;13) | 44.0 [18.3 to 105.9] | 5.1 [3.1 to 8.6] | 83.5 [16.2 to 431.7] | 9.5 [4.3 to 21.2]

3. Primary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above Pre-defined Cut-off Values Enzyme-Linked Immunosorbent Assay (ELISA).
Description: Anti-hepatitis B surface antigen (anti-HBs) antibody cut-off values assessed include 1.0 and 10 mIU/mL.
Time Frame: At Years 15, 16, 17, 18, 19 and 20
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Number analyzed (Participants) | 17 | 15 | 12 | 17
subjects
  Year 15 (≥ 1.0 mIU/mL) (N=17;15;12;17) | 17 | 7 | 10 | 11
  Year 15 (≥ 10 mIU/mL) (N=17;15;12;17) | 16 | 4 | 9 | 7
  Year 16 (≥ 1.0 mIU/mL) (N=15;13;12;16) | 15 | 9 | 12 | 11
  Year 16 (≥ 10 mIU/mL) (N=15;13;12;16) | 14 | 6 | 10 | 8
  Year 17 (≥ 1.0 mIU/mL) (N=17;13;11;13) | 15 | 7 | 11 | 10
  Year 17 (≥ 10 mIU/mL) (N=17;13;11;13) | 15 | 2 | 9 | 5
  Year 18 (≥ 1.0 mIU/mL) (N=14;14;10;13) | 14 | 7 | 10 | 8
  Year 18 (≥ 10 mIU/mL) (N=14;14;10;13) | 13 | 3 | 7 | 7
  Year 19 (≥ 1.0 mIU/mL) (N=14;12;8;11) | 13 | 7 | 8 | 8
  Year 19 (≥ 10 mIU/mL) (N=14;12;8;11) | 12 | 3 | 6 | 6
  Year 20 (≥ 1.0 mIU/mL) (N=13;13;6;12) | 13 | 9 | 5 | 10
  Year 20 (≥ 10 mIU/mL) (N=13;13;6;12) | 11 | 5 | 5 | 6

4. Primary Outcome: Adjusted Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above Pre-defined Cut-off Values as Measured by ChemiLuminescence ImmunoAssay (CLIA)
Description: Anti-hepatitis B surface antigen (anti-HBs) antibody cut-off values assessed include 1.0 and 10 mIU/mL.
  Note: Missing CLIA anti-HBs concentrations, for subjects with ELISA results available, are estimated by multiple imputations and GMCs and number of subjects were adjusted for these imputations.
Time Frame: At Years 19 and 20
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | ENGERIX 4D + HBIG GROUP | ENGERIX 3D + HBIG GROUP | ENGERIX 4D | ENGERIX 3D GROUP
Number analyzed (Participants) | 16 | 13 | 7 | 13
Subjects
  Year 19 (≥ 1.0 mIU/mL) (N=14;12;6;11) | 13.0 | 4.2 | 6.0 | 7.0
  Year 19 (≥ 10 mIU/mL) (N=14;12;6;11) | 12.0 | 3.9 | 5.0 | 4.0
  Year 20 (≥ 1.0 mIU/mL) (N=16;13;7;13) | 13.1 | 5.4 | 6.0 | 6.3
  Year 20 (≥ 10 mIU/mL) (N=16;13;7;13) | 12.2 | 2.1 | 5.0 | 5.8

5. Primary Outcome: Number of Subjects With Positive Results for Serological Markers for Hepatitis B Infection
Description: Serological markers for hepatitis B infection assessed are hepatitis B surface antigen (HBsAg), antibodies to hepatitis B core antigen (anti-HBc), hepatitis B e antigen (HBeAg) and antibodies to hepatitis B e antigen (anti-HBe).
Time Frame: At Years 15, 16, 17, 18, 19 and 20
Population: Analysis was performed on the Long Term Total Cohort (LT total cohort) on subjects with available data for the specified marker.
Measure: Number; unit: subjects
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Number analyzed (Participants) | 19 | 19 | 16 | 22
subjects
  Year 15 HBsAg (N=19;19;14;21) | 0 | 1 | 0 | 3
  Year 15 Anti-HBc (N=19;19;14;21) | 4 | 7 | 1 | 9
  Year 15 HBeAg (N=4;7;1;8) | 0 | 1 | 0 | 1
  Year 15 Anti-HBe (N=4;7;1;8) | 1 | 1 | 0 | 3
  Year 16 HBsAg (N=16;17;16;22) | 2 | 0 | 2 | 5
  Year 16 Anti-HBc (N=16;17;16;22) | 4 | 5 | 1 | 9
  Year 16 HBeAg (N=6;5;3;11) | 1 | 1 | 0 | 3
  Year 16 Anti-HBe (N=6;5;3;11) | 0 | 1 | 0 | 2
  Year 17 HBsAg (N=19;17;13;19) | 6 | 0 | 3 | 6
  Year 17 Anti-HBc (N=19;17;13;20) | 5 | 5 | 1 | 8
  Year 17 HBeAg (N=9;5;4;10) | 0 | 0 | 0 | 1
  Year 17 Anti-HBe (N=9;5;4;10) | 1 | 0 | 0 | 3
  Year 18 HBsAg (N=16;17;14;20) | 3 | 1 | 3 | 5
  Year 18 Anti-HBc (N=16;17;14;20) | 5 | 6 | 1 | 8
  Year 18 HBeAg (N=8;7;4;10) | 0 | 0 | 0 | 1
  Year 18 Anti-HBe (N=8;7;4;10) | 1 | 1 | 0 | 2
  Year 19 HBsAg (N=17;16;12;18) | 4 | 3 | 3 | 5
  Year 19 Anti-HBc (N=17;16;12;18) | 4 | 5 | 2 | 9
  Year 19 HBeAg (N=8;7;5;10) | 0 | 0 | 0 | 2
  Year 19 Anti-HBe (N=8;7;5;10) | 1 | 1 | 0 | 3
  Year 20 HBsAg (N=19;17;12;20) | 6 | 5 | 4 | 12
  Year 20 Anti-HBc (N=19;17;12;20) | 5 | 7 | 2 | 8
  Year 20 HBeAg (N=8;7;6;14) | 1 | 0 | 0 | 1
  Year 20 Anti-HBe (N=10;9;6;15) | 1 | 0 | 0 | 3

6. Primary Outcome: Number of Subjects With Different Hepatitis B Infection Statuses
Description: Categories hepatitis B (HB) infection:
  1. Chronic infection: HBsAg and anti-HBc pos (pos) in more than two consecutive samples
  2. False positive: single HB marker (HBsAg, HBeAg, anti-HBc) pos + all other markers negative (neg) in one sample. Consecutive time points all neg.
  3. Possible subclinical breakthrough infection: One or more HB markers pos in one or more consecutive samples.
  4. Isolated natural booster: >4-fold increase of anti-HBs concentrations if <100 mIU/mL at previous sample OR >2- fold increase of anti-HBs concentrations if >=100 mIU/mL at previous sample + other markers neg
Time Frame: Over the entire follow up period (Final assessment of clinical significance was analyzed after the Year 20 time point)
Population: Analysis was performed on the Long Term Total Cohort (LT total cohort). The maximum amount of subjects who have participated in any of the time points in this study has been given as number of participants analyzed.
Measure: Number; unit: subjects
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Number analyzed (Participants) | 19 | 19 | 16 | 22
subjects
  Chronic HB infection | 0 | 0 | 0 | 4
  False positive | 5 | 5 | 9 | 10
  Possible subclinical breakthrough HB infection | 9 | 12 | 4 | 10
  Isolated natural booster | 8 | 8 | 9 | 7

ADVERSE EVENTS:
Description: As no adverse events data were collected during this study the number of participants at risk is 0 for all groups.
Arm/Group | Engerix 4D + HBIg Group | Engerix 3D + HBIg Group | Engerix 4D | Engerix 3D Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). Additional tables have been generated following partial retesting and reanalysis of the results at Years 19 and 20.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.